CLINICAL TRIAL: NCT05971095
Title: Percutaneous Femoral Nerve Neuromodulation for Postoperative Analgesia and Functional Recovery Following Knee Arthroplasty.
Brief Title: Comparison Between Percutaneous Femoral Nerve Neuromodulation Associated With Femoral Nerve Block and Standard Clinical Practice in Patients Undergoing Knee Arthroplasty.
Acronym: NEPFAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital General Universitario de Valencia (Other)
Responsible Party: Principal Investigator, FERRAN MARQUES PEIRO, Principal Investigator, Hospital General Universitario de Valencia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20121994
Record Dates: First submitted 2023-07-06; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Acute Pain
Keywords: PENS; Neuromodulation; Percutaneous peripheral nere stimulation; Postoperative pain; Acute pain after surgery; Total Knee arthtolasty
MeSH Terms: conditions — Acute Pain; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: This is an analytical study (with hypothesis testing) of a single-center, unblinded, randomized clinical trial. The patients will be separated between the intervention group and the control group.
  To carry out the assignment of interventions, a methodology by blocks of 2 without stratification will be used. To obtain the sequence of random numbers, the official Clinical Trial Randomization Tool of the National Cancer Institute (USA) will be used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Neuromodulation group (Experimental): The maximum isometric contraction force of the quadriceps will be measured prior to the neuromodulation program using a hand dynamometer.
  The percutaneous neuromodulation program will begin using the EPTE® Bipolar System device. The two stimulation protocols will be applied consecutively. Firstly, the high-frequency protocol (HFS) will be applied using the pulsed square waveform and 5 bursts of stimulation lasting 5 seconds at a frequency of 100 Hz separated by 55 s interval between bursts.
  The low-frequency protocol (LFS) with stimulation at 2 Hz for 16 min with an intensity of 1000μA will subsequently be switched to.
  The surgical intervention will be carried out by subarachnoid block with local anesthetic in accordance with the usual practice.
  After its completion, a single injection block of the femoral nerve will be performed with a long-acting local anesthetic , a regional anesthesia technique included in routine clinical practice.
  Interventions: Device: Percutaneous neuromodulation using the EPTE® Bipolar System device
- Control group (No Intervention): The neuromodulation program will not be carried out. Only the maximum contraction force of the quadriceps prior to subarachnoid block will be measured. After the intervention, the femoral nerve block will be performed following the usual clinical practice.

INTERVENTIONS:
Device: Percutaneous neuromodulation using the EPTE® Bipolar System device — The two stimulation protocols will be applied consecutively. Firstly, the high-frequency protocol (HFS) will be applied in order to produce potentiation of the non-nociceptive pathway, using the pulsed square waveform and 5 bursts of stimulation lasting 5 seconds at a frequency of 100 Hz separated by 55 s interval between bursts. Adjustments to amplitude and pulse width are made until the patient experiences paresthesias at a perceptible but not painful intensity, and the intensity will be set 200 μA above the detection threshold for each subject.
  In order to depress the nociceptive pathway, the low-frequency protocol (LFS) with stimulation at 2 Hz for 16 min with an intensity of 1000μA will subsequently be switched to. To ensure the recruitment of higher threshold type C nociceptive fibers, the intensity level will be programmed at the pain threshold for each subject.
  Arms: Neuromodulation group

SUMMARY:
The goal of this clinical trial is to compare the maximum isometric contraction force differential of the quadriceps in the postoperative period after the use of a peripheral nerve neuromodulation program in patients undergoing knee arthroplasty. The main questions it aims to answer are if the combination of a peripheral neuromodulation program in the perioperative period improves analgesic quality and short-term functional recovery in patients undergoing knee arthroplasty,

Participants will be asked to reach a maximum knee extension prior to neurostimulation Patients will have the electrodes inserted under direct ultrasound vision and placed near the femoral nerve.

Researchers will compare whether there is a difference in both quadriceps contraction force and analgesia between the stimulated group and the control group.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years
* Those who sign the informed consent
* Not pregnant
* Cognitive capacity that allows subjective postoperative evaluations.

Exclusion Criteria:

* Under 18 years old
* IC rejection or withdrawal
* Pregnancy
* Cognitive impairment
* Contraindication for Regional Anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Quadriceps maximal isometric contraction force differential after the use of a peripheral nerve neuromodulation program with direct current at low frequency combined with high frequency | Before neuromodulation, immediately after the first phase of the program, and 24 hours after it.
  To compare (analyze) the differential of the maximum isometric contraction force of the quadriceps in the postoperative period after the use of a peripheral nerve neuromodulation program with direct current at low frequency combined with high frequency compared to the usual practice.

SECONDARY OUTCOMES:
VAS score and Opioid use | In the immediate postoperative period in the PACU and at 24 hours
  To compare the analgesic efficacy with the use of the described neuromodulation program versus the usual practice, in which it is not performed, in patients undergoing knee arthroplasty.

CONTACTS AND LOCATIONS:
Overall Officials: JOSE DE ANDRES IBAÑEZ, FEA, Study Director — CONSORCIO HOSPITAL GENERAL DE VALENCIA
Locations (1):
- Hospital General Universitario de Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ripolles-Melchor J, Abad-Motos A, Diez-Remesal Y, Aseguinolaza-Pagola M, Padin-Barreiro L, Sanchez-Martin R, Logrono-Egea M, Catala-Bauset JC, Garcia-Orallo S, Bisbe E, Martin N, Suarez-de-la-Rica A, Cuellar-Martinez AB, Gil-Trujillo S, Estupinan-Jimenez JC, Villanova-Baraza M, Gil-Lapetra C, Perez-Sanchez P, Rodriguez-Garcia N, Ramiro-Ruiz A, Farre-Tebar C, Martinez-Garcia A, Arauzo-Perez P, Garcia-Perez C, Abad-Gurumeta A, Minambres-Villar MA, Sanchez-Campos A, Jimenez-Lopez I, Tena-Guerrero JM, Marin-Pena O, Sanchez-Merchante M, Vicente-Gutierrez U, Cassinello-Ogea MC, Ferrando-Ortola C, Berges-Gutierrez H, Fernanz-Anton J, Gomez-Rios MA, Bordonaba-Bosque D, Ramirez-Rodriguez JM, Garcia-Erce JA, Aldecoa C; Postoperative Outcomes Within Enhanced Recovery After Surgery Protocol in Elective Total Hip and Knee Arthroplasty (POWER2) Study Investigators Group for the Spanish Perioperative Audit and Research Network (REDGERM). Association Between Use of Enhanced Recovery After Surgery Protocol and Postoperative Complications in Total Hip and Knee Arthroplasty in the Postoperative Outcomes Within Enhanced Recovery After Surgery Protocol in Elective Total Hip and Knee Arthroplasty Study (POWER2). JAMA Surg. 2020 Apr 1;155(4):e196024. doi: 10.1001/jamasurg.2019.6024. Epub 2020 Apr 15. PMID 32049352
- [Background] Dos'Santos T, Thomas C, Comfort P, McMahon JJ, Jones PA. Relationships between Isometric Force-Time Characteristics and Dynamic Performance. Sports (Basel). 2017 Sep 13;5(3):68. doi: 10.3390/sports5030068. PMID 29910428
- [Background] Maffiuletti NA. Assessment of hip and knee muscle function in orthopaedic practice and research. J Bone Joint Surg Am. 2010 Jan;92(1):220-9. doi: 10.2106/JBJS.I.00305. PMID 20048117
- [Background] Rice DA, McNair PJ. Quadriceps arthrogenic muscle inhibition: neural mechanisms and treatment perspectives. Semin Arthritis Rheum. 2010 Dec;40(3):250-66. doi: 10.1016/j.semarthrit.2009.10.001. Epub 2009 Dec 2. PMID 19954822
- [Result] Ma HH, Chou TA, Tsai SW, Chen CF, Wu PK, Chen WM. The efficacy of continuous versus single-injection femoral nerve block in Total knee Arthroplasty: a systematic review and meta-analysis. BMC Musculoskelet Disord. 2020 Feb 24;21(1):121. doi: 10.1186/s12891-020-3148-1. PMID 32093655
- [Result] Hussain N, Ferreri TG, Prusick PJ, Banfield L, Long B, Prusick VR, Bhandari M. Adductor Canal Block Versus Femoral Canal Block for Total Knee Arthroplasty: A Meta-Analysis: What Does the Evidence Suggest? Reg Anesth Pain Med. 2016 May-Jun;41(3):314-20. doi: 10.1097/AAP.0000000000000376. No abstract available. PMID 27035459
- [Result] Angers M, Belzile EL, Vachon J, Beauchamp-Chalifour P, Pelet S. Negative Influence of femoral nerve block on quadriceps strength recovery following total knee replacement: A prospective randomized trial. Orthop Traumatol Surg Res. 2019 Jun;105(4):633-637. doi: 10.1016/j.otsr.2019.03.002. Epub 2019 Mar 28. PMID 30928275
- [Result] Gilmore C, Ilfeld B, Rosenow J, Li S, Desai M, Hunter C, Rauck R, Kapural L, Nader A, Mak J, Cohen S, Crosby N, Boggs J. Percutaneous peripheral nerve stimulation for the treatment of chronic neuropathic postamputation pain: a multicenter, randomized, placebo-controlled trial. Reg Anesth Pain Med. 2019 Jun;44(6):637-645. doi: 10.1136/rapm-2018-100109. Epub 2019 Apr 5. PMID 30954936
- [Result] Plaza-Manzano G, Gomez-Chiguano GF, Cleland JA, Arias-Buria JL, Fernandez-de-Las-Penas C, Navarro-Santana MJ. Effectiveness of percutaneous electrical nerve stimulation for musculoskeletal pain: A systematic review and meta-analysis. Eur J Pain. 2020 Jul;24(6):1023-1044. doi: 10.1002/ejp.1559. Epub 2020 Apr 4. PMID 32171035
- [Result] Strand NH, D'Souza R, Wie C, Covington S, Maita M, Freeman J, Maloney J. Mechanism of Action of Peripheral Nerve Stimulation. Curr Pain Headache Rep. 2021 May 11;25(7):47. doi: 10.1007/s11916-021-00962-3. PMID 33973135
- [Result] Klein T, Magerl W, Hopf HC, Sandkuhler J, Treede RD. Perceptual correlates of nociceptive long-term potentiation and long-term depression in humans. J Neurosci. 2004 Jan 28;24(4):964-71. doi: 10.1523/JNEUROSCI.1222-03.2004. PMID 14749441
- [Result] Beltra P, Ruiz-Del-Portal I, Ortega FJ, Valdesuso R, Delicado-Miralles M, Velasco E. Sensorimotor effects of plasticity-inducing percutaneous peripheral nerve stimulation protocols: a blinded, randomized clinical trial. Eur J Pain. 2022 May;26(5):1039-1055. doi: 10.1002/ejp.1928. Epub 2022 Mar 3. PMID 35191131
- [Result] Ilfeld BM, Plunkett A, Vijjeswarapu AM, Hackworth R, Dhanjal S, Turan A, Cohen SP, Eisenach JC, Griffith S, Hanling S, Sessler DI, Mascha EJ, Yang D, Boggs JW, Wongsarnpigoon A, Gelfand H; PAINfRE Investigators. Percutaneous Peripheral Nerve Stimulation (Neuromodulation) for Postoperative Pain: A Randomized, Sham-controlled Pilot Study. Anesthesiology. 2021 Jul 1;135(1):95-110. doi: 10.1097/ALN.0000000000003776. PMID 33856424
- [Result] Gallego-Sendarrubias GM, Arias-Buria JL, Ubeda-D'Ocasar E, Hervas-Perez JP, Rubio-Palomino MA, Fernandez-de-Las-Penas C, Valera-Calero JA. Effects of Percutaneous Electrical Nerve Stimulation on Countermovement Jump and Squat Performance Speed in Male Soccer Players: A Pilot Randomized Clinical Trial. J Clin Med. 2021 Feb 10;10(4):690. doi: 10.3390/jcm10040690. PMID 33578911